CLINICAL TRIAL: NCT02060981
Title: Primary Medication Adherence Phase 2 Evaluation of a Decision Support Tool
Brief Title: Evaluation of a Decision Support Tool
Acronym: PRIMA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Foundation for Informed Medical Decision Making (Other)
Responsible Party: Principal Investigator, Jennifer Polinski, Assistant Professor and Epidemiologist, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-P-00008959; #2013P001295/BWH (Other: Partners IRB)
Record Dates: First submitted 2014-02-10; First posted 2014-02-12 (Estimated); Last update posted 2015-02-18 (Estimated); Status verified 2015-02

CONDITIONS: Medication Adherence; Hypertension; Decision Making, Shared; Patient-Centered Outcomes Research
Keywords: Randomized controlled trial; Primary medication adherence; Decision-support tool; Patient-centered outcomes research; Antihypertensive medications; One-on-one patient interviews
MeSH Terms: conditions — Medication Adherence; Hypertension | interventions — Interviews as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Interview only (Active Comparator): Patients will be asked to participate in an interview regarding their views on hypertension and taking medications to treat hypertension.
  Interventions: Behavioral: Interview Only
- Control (Placebo Comparator): Control group patients will then be mailed an American Heart Association brochure regarding hypertension and a brief, 5-question, paper-based survey. These patients will be asked to review the brochure, complete the survey, and mail it back to the research team using a self-addressed stamped envelope.
  Interventions: Behavioral: Control
- Interview plus decision support tool (Experimental): Patients will be asked to participate in an interview regarding their views on hypertension and taking medications to treat hypertension, and to provide feedback regarding a new tool for helping patients learn more about their medications. Interview plus patients' index date for follow-up is the date of the scheduled interview.
  Interventions: Behavioral: Interview plus decision support tool

INTERVENTIONS:
Behavioral: Control — Control group patients will then be mailed an American Heart Association brochure regarding hypertension and a brief, 5-question, paper-based survey.
  Arms: Control
Behavioral: Interview Only — Patients will be asked to participate in an interview regarding their views on hypertension and taking medications to treat hypertension.
  Arms: Interview only
Behavioral: Interview plus decision support tool — Patients will be asked to participate in an interview regarding their views on hypertension and taking medications to treat hypertension and to provide feedback regarding a new decision support tool for helping patients learn more about their medications.
  Arms: Interview plus decision support tool

SUMMARY:
Investigators will conduct a randomized trial with patients, through one-on-one interviews, to evaluate their understanding of and willingness to use a decision support tool and to determine if receiving and discussing the decision support tool improves the likelihood that a patient is adherent to a new antihypertensive medication.

ELIGIBILITY:
Inclusion Criteria:

* does not pick up a prescription for a new antihypertensive medication within 14 days as identified by CVS pharmacy, their retail pharmacy provider.
* High blood pressure diagnosis

Exclusion Criteria:

* under age 25.

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-03 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of antihypertensive medication fills | 6 months
  The proportion of patients in each group who picked up a prescription for an antihypertensive medication in any class during the follow-up period. Investigators will calculate cumulative incidences among all patients, whether or not they successfully completed the interview or returned the paper-based survey (Intention to Treat) and among only those patients who did complete the interview or returned the paper-based survey (As Treated).

SECONDARY OUTCOMES:
Patient Interviews | 5 months
  One-on-one structured interviews will ask about participants' preferences, attitudes and beliefs regarding primary adherence and/or use of a decision support tool.

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Polinski, Sc.D., Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States